CLINICAL TRIAL: NCT02416323
Title: Effectiveness and Implementation of a Mental Health Intervention for ASD
Acronym: AIM HI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lauren Brookman-Frazee, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2011-4131; R01MH094317 (NIH)
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Community therapist delivers routine care to participant child with no training in AIM HI.
- AIM HI Training (Other): Therapist enrolls in AIM HI training
  Interventions: Other: AIM HI Training

INTERVENTIONS:
Other: AIM HI Training
  Arms: AIM HI Training

SUMMARY:
The purpose of this study is to test the effectiveness of training community mental health therapists to deliver a mental health intervention for ASD ("AIM HI") and study the process of implementing AIM HI in community mental health programs.

DETAILED DESCRIPTION:
This study is a randomized controlled effectiveness trial of AIM HI ("An Individualized Mental Health Intervention for ASD"), an intervention designed specifically for implementation in community mental health clinics, to reduce problem behavior among school-age children with autism spectrum disorders (ASD). Although the individual components of AIM HI are well-established evidence-based practice strategies and pilot study data indicate that child behavior problems decrease when their community mental health therapists deliver AIM HI, the effectiveness of the protocol has not been established. Therefore, the primary aims are to test the impact of training community therapists in AIM HI on child and family outcomes and determine how child/ family characteristics and level of therapist fidelity moderate treatment effects. The secondary aim is to collect initial data on implementation outcomes and conduct exploratory analyses to identify barriers and facilitators of AIM HI implementation (e.g., intervention, organization, provider characteristics). This study has the potential to make a significant impact by building local capacity to serve school-age children with ASD in routine service settings, and advancing the science on the effectiveness of packaging evidence-based practices (EBPs) for specific services settings. It will also produce generalizable knowledge about implementation that can be applied for this population/ setting.

ELIGIBILITY:
Inclusion Criteria for Therapists

1. Employed as staff or a trainee at participating clinic (publicly-funded mental health program)
2. Employed for at least the next 7 months (i.e., practicum or internship not ending in next 7 months).
3. Has an eligible client on current caseload (see below).

Inclusion Criteria for Child/ Parent Participants

1. Child age 5-13 years.
2. Has a current ASD diagnosis on record.
3. Meets criteria for ASD on the Autism Diagnostic Observation Schedule (ADOS) or exhibits other clinical indicators of ASD
4. English or Spanish speaking.

Exclusion Criteria for Child/ Parent Participants

1. Child does not present with challenging behaviors.
2. Child does not meet criteria for ASD on the ADOS or exhibit other clinical indicators of ASD

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 609 (Actual)
Dates: Start 2012-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change since baseline in child behaviors on the Eyberg Child Behavior Inventory (ECBI) | Study Enrollment, 6, 12, 18 months post study enrollment

SECONDARY OUTCOMES:
Change since baseline in child behaviors on the Social Skills Improvement System (SSIS) Competing Behavior Scale | Study Enrollment, 6, 12, 18 months post study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Services Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Caplan B, Chlebowski C, Lind T, Rangel E, Brookman-Frazee L. Therapist-Reported Adaptations to an Autism Intervention: Family-Level Predictors and Associations with Fidelity. J Autism Dev Disord. 2024 Oct 28. doi: 10.1007/s10803-024-06603-z. Online ahead of print. PMID 39466584
- [Derived] Caplan B, Lind T, Chlebowski C, Martinez K, May GC, Gomez Alvarado CJ, Brookman-Frazee L. Training Community Therapists in AIM HI: Individual Family and Neighborhood Factors and Child/Caregiver Outcomes. J Clin Child Adolesc Psychol. 2024 Sep-Oct;53(5):783-795. doi: 10.1080/15374416.2022.2096046. Epub 2022 Jul 26. PMID 35881774
- [Derived] Brookman-Frazee L, Chlebowski C, Villodas M, Roesch S, Martinez K. Training Community Therapists to Deliver an Individualized Mental Health Intervention for Autism Spectrum Disorder: Changes in Caregiver Outcomes and Mediating Role on Child Outcomes. J Am Acad Child Adolesc Psychiatry. 2021 Mar;60(3):355-366. doi: 10.1016/j.jaac.2020.07.896. Epub 2020 Aug 2. PMID 32755632
- [Derived] Brookman-Frazee L, Roesch S, Chlebowski C, Baker-Ericzen M, Ganger W. Effectiveness of Training Therapists to Deliver An Individualized Mental Health Intervention for Children With ASD in Publicly Funded Mental Health Services: A Cluster Randomized Clinical Trial. JAMA Psychiatry. 2019 Jun 1;76(6):574-583. doi: 10.1001/jamapsychiatry.2019.0011. PMID 30840040
- [Derived] Stadnick N, Chlebowski C, Baker-Ericzen M, Dyson M, Garland A, Brookman-Frazee L. Psychiatric comorbidity in autism spectrum disorder: Correspondence between mental health clinician report and structured parent interview. Autism. 2017 Oct;21(7):841-851. doi: 10.1177/1362361316654083. Epub 2016 Jul 11. PMID 27407039